CLINICAL TRIAL: NCT03844594
Title: Safety and Efficacy of Eptifibatide in Endovascular Treatment of Acute Ischemic Stroke: a Single-arm, Open-label, Multicenter Clinical Trial
Brief Title: Eptifibatide in Endovascular Treatment of Acute Ischemic Stroke (EPOCH)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Zhongrong Miao, Chief of Department of Neurological Intervention, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019EPOCH19011912
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Eptifibatide; Endovascular Treatment; Recovery of Dysfunction
MeSH Terms: conditions — Ischemic Stroke | interventions — Eptifibatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eptifibatide Drug: Eptifibatide Injection (Experimental)
  Interventions: Drug: Eptifibatide Injection

INTERVENTIONS:
Drug: Eptifibatide Injection — Recommendation: first, intravenously or intraductal injection of 135ug / kg (completed in 5 minutes), followed by continuous intravenous infusion of 0.75ug / kg / min for 24 hours.

SUMMARY:
The study is a single-arm, open-label, multicenter clinical trial.The primary purpose of this trial is to evaluate the incidence of symptomatic intracranial hemorrhage in patients with acute ischemic stroke within 48 hours after the use of Eptifibatide injection. Patients with acute ischemic stroke treated with intravascular thrombolytic therapy, mechanical thrombolysis, angioplasty and so on were treated with Eptifibatide injection on the first day, followed by the second day, the third day, the discharge day and the 90 days.

DETAILED DESCRIPTION:
The study is a single-arm, open-label, multicenter clinical trial.A total of 220 patients (Age≥18years) with acute ischemic stroke treated with intravascular thrombolysis, mechanical thrombolysis, angioplasty, etc., were treated with Eptifibatide, providing informed consent and medication.The recommended dose of this study was: first, 135ug / kg was injected intravenously or intraductal (within 5 minutes), followed by continuous intravenous infusion of 0.75 ug / kg / min for 24 h. In special cases, it is up to the operator to decide whether to reinject or increase the dosage according to experience. The maximum dose for the first time was 180ug / kg, if necessary, with a 10-minute interval of intravenously or intraductal injection, and a maximum dose of 180ug / kg, intravenously / intraductal injection of no more than 360ug / kg. Continuous intravenous infusion does not exceed 2ug/kg/ Min. Then the second day, the third day, the discharge and 90 days visit. Follow-up information included vital signs and physical examination, observation of symptomatic intracranial hemorrhage, NIHSS scale, and recording of current drug use by AE,SAE.The trial is anticipated to last from January 2019 to December 2019 with 220 subjects recruited form 15 centers in China. All the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese GCP standard. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by Institutional Review Board (IRB) and Ethics Committee(EC) in Being Tiantan hospital, Capital Medical University.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years.
2. Acute ischemic stroke.
3. Treated with endovascular treatment, including intra-arterial thrombolysis, mechanical thrombectomy, and angioplasty.
4. Written informed consent obtained from patient or patient's legally authorized representative.

Exclusion Criteria:

1. Failed to vascular recanalization (mTICI≤1).
2. Diagnosis of intracranial hemorrhagic disease, such as intracranial hemorrhage, subarachnoid hemorrhage and so on.
3. Known coagulopathy, Systemic Bleeding Tendency, or baseline platelet count < 100000/mm3.
4. History of chronic hepatopathy, liver and kidney dysfunction, elevating ALT (> 3 times normal upper limit), elevating serum creatinine (> 2 times normal upper limit).
5. Patients with severe hypertension (systolic blood pressure > 200mmHg or diastolic blood pressure > 110mmHg).
6. Known drug or food allergy.
7. Used other Glycoprotein IIb/IIIa receptor antagonists.
8. Contraindications for DSA, severe contrast media allergy or iodine contrast media absolute contraindications.
9. Childbearing age women whose pregnancy tests were negative refused to take effective contraception. Pregnant or lactating or positive pregnancy test on admission.
10. Incapable to follow this study for mental illness, cognitive or emotional disorder.
11. The researchers do not consider the participants appropriate to get into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-04-06 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptomatic intracranial hemorrhage | Within 48 hours
  Incidence of symptomatic Intracranial Hemorrhage within 48 hours after treatment

SECONDARY OUTCOMES:
Cerebral parenchymal hemorrhage type (PH1) and (PH2) | 48 hours
  The incidence of cerebral parenchymal hemorrhage type (PH1) and (PH2) for 48 hours of treatment
Serious adverse events | Within 48 hours
  Proportion of serious adverse events occurring within 48 hours of treatment
Total death rate | Within 48 hours
  Total death rate within 48 hours of treatment
Adverse events | Within 48 hours
  Proportion of adverse events within 48 hours of treatment
Serious adverse events | Within 90 days
  Proportion of serious adverse events within 90 days of treatment
Total death rate | Within 90 days
  Total death rate within 90 days of treatment
Adverse events | Within 90 days
  Proportion of adverse events treated within 90 days
Vascular recanalization | 24 hours
  Proportion of vascular recanalization at the first 24 hours during the therapy
Favorable clinical outcomes | 90 days
  Proportion of patients achieve favorable clinical outcomes (mRS 0-2) after 90 days of treatment
Neurological recovery | 90 days
  The recovery of neurological deficits assessed by the difference of the 90 days NIHSS to the baseline NIHSS
Recurrent ischemic stroke | 90 days
  Proportion of recurrent ischemic stroke after 90 days of treatment
Combined vascular events | 90 days
  Proportion of combined vascular events (recurrent ischemic stroke, myocardial infarction and vascular death) at 90 days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ma G, Sun X, Cheng H, Burgin WS, Luo W, Jia W, Liu Y, He W, Geng X, Zhu L, Chen X, Shi H, Xu H, Zhang L, Wang A, Mo D, Ma N, Gao F, Song L, Huo X, Deng Y, Liu L, Luo G, Jia B, Tong X, Liu L, Ren Z, Miao Z; EPOCH Study and ANGEL-ACT Study Groups. Combined Approach to Eptifibatide and Thrombectomy in Acute Ischemic Stroke Because of Large Vessel Occlusion: A Matched-Control Analysis. Stroke. 2022 May;53(5):1580-1588. doi: 10.1161/STROKEAHA.121.036754. Epub 2022 Feb 2. PMID 35105182